CLINICAL TRIAL: NCT00067925
Title: Incorporating More Physical Activity and Calcium in Teens (IMPACT): A School-Based Osteoporosis Prevention Program for Adolescent Girls
Brief Title: A School-Based Osteoporosis Prevention Program for Adolescent Girls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037767 (NIH)
Record Dates: First submitted 2003-09-03; First posted 2003-09-04 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2003-08

CONDITIONS: Osteoporosis
Keywords: Weight-bearing physical activity; Calcium intake; School-based health education; Adolescent girls; Child nutrition; Diet
MeSH Terms: conditions — Osteoporosis | interventions — Calcium

INTERVENTIONS:
Behavioral: Incorporating More Physical Activity and Calcium in Teens (IMPACT) Program

SUMMARY:
The Incorporating More Physical Activity and Calcium in Teens (IMPACT) study was a behaviorally-based middle school nutrition and physical activity program for the prevention of osteoporosis. The goal of IMPACT was to increase calcium intake and physical activity to help build bone mass in girls.

DETAILED DESCRIPTION:
Peak bone mass is achieved during the first twenty years of life, and dietary and activity patterns that contribute to the formation of peak bone mass are developed during childhood. The IMPACT intervention was designed to increase bone density and ultimately prevent osteoporosis during adulthood. IMPACT included physical education, food service, and classroom environmental and behavioral components and was delivered by physical education (PE) specialists, food service personnel, and classroom teachers.

A group of 718 sixth grade girls (mean age 11.1) from twelve middle schools in central Texas participated in the study. The group was 72% non-Hispanic white, 12% Hispanic, 5% African American, and 11% other ethnicity. After baseline measurements were completed in the fall of 2000, the twelve middle schools were pair-matched based on school characteristics (ethnicity, % economically disadvantaged, % girls in athletics) to a control (usual health education program) or the IMPACT program. The intervention was implemented for 18 months and consisted of three major components: a PE component, which emphasized daily weight-bearing activities (WBA); a health lessons component consisting of sixteen behaviorally-based lessons which emphasized WBA, calcium-rich foods, and osteoporosis prevention; and a food service component.

Outcome measures included physical properties of the students' heel bones, calcium consumption, physical activity, and psychosocial factors believed to be precursors to these behaviors. Changes at the school environmental level, such as the number of calcium rich foods offered in the cafeteria and the number of opportunities offered for weight-bearing and aerobic activity, were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Girls enrolled in 6th grade of selected schools
* Student assent
* Parental consent
* No fractures or medications that compromise bone health or strength
* Enrolled in 2 semesters of physical education

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 718
Dates: Start 2000-09; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Deanna M Hoelscher, PhD, Principal Investigator — University of Texas-Houston School of Public Health

REFERENCES:
- [Derived] Sharma SV, Hoelscher DM, Kelder SH, Diamond P, Day RS, Hergenroeder A. Psychosocial factors influencing calcium intake and bone quality in middle school girls. J Am Diet Assoc. 2010 Jun;110(6):932-6. doi: 10.1016/j.jada.2010.03.013. PMID 20497785
- [Derived] Sharma SV, Hoelscher DM, Kelder SH, Diamond PM, Day RS, Hergenroeder AC. A path analysis to identify the psychosocial factors influencing physical activity and bone health in middle-school girls. J Phys Act Health. 2009 Sep;6(5):606-16. doi: 10.1123/jpah.6.5.606. PMID 19953837
- [Derived] Sharma SV, Hoelscher DM, Kelder SH, Day RS, Hergenroeder A. Psychosocial, environmental and behavioral factors associated with bone health in middle-school girls. Health Educ Res. 2009 Apr;24(2):173-84. doi: 10.1093/her/cyn009. Epub 2008 Mar 21. PMID 18359949